CLINICAL TRIAL: NCT05713344
Title: Evaluation of Pain Phenotypes in Chronic Pancreatitis and Identification of Clinical Surrogates of Pancreatic Neuropathy
Brief Title: Pain Phenotypes in Chronic Pancreatitis
Acronym: PIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Collaborators: All India Institute of Medical Sciences (Other); SIDS Hospital and Research Center, Surat (Unknown); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Rupjyoti Talukdar, Director, Pancreatology; Head, Pancreas Research Group and Division of Gut Microbiome Research, Asian Institute of Gastroenterology, India
Other Study IDs: PIPver01
Record Dates: First submitted 2023-01-22; First posted 2023-02-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical history — Detailed clinical history including demographic details, pain details (character, pattern, location, change in character, involvement of new areas), duration of disease, co-morbidities, family history, adverse life events, sleep details, details of stress/anxiety.
Other: Clinical examination — Thorough clinical examination, anthropometric measurement, assessment of pain (Izbicki score, Visual analog scale, modified brief pain inventory, pain catastrophising score, painDetect)
Other: Evaluation of quality of life — Use of the EORTC QLQ c30 with PAN 28 to evaluate quality of life
Other: Evaluation of mental state — Use of Beck depression inventory and Hospital Anxiety Depression score to evaluate depression and anxiety
Diagnostic Test: Pancreatic quantitative sensory testing — Pancreatic quantitative sensory testing will be performed to evaluate temporal summation, pain detection threshold, pain tolerance threshold, and conditioned pain modulation.

SUMMARY:
Chronic pancreatitis (CP) is characterised by recurrent abdominal pain. The pathological hallmarks of CP is pancreatic stellate cell activation that results in persistent inflammation and progressive fibrosis. It has been shown in various clinical and experimental studies that with disease progression there could be pancreatic neural inflammation, spinal sensitization and eventually alteration in the pain modulating architecture within the brain (widespread sensitization). These events result in different types of pain (nociceptive and neuropathic) in patients with CP, which may dynamically change during disease progression.

Since the treatment for different mechanisms are unique, it becomes important to identify the predominant type of pain. Recently, pancreatic quantitative sensory testing (P-QST) has emerged as a valuable tool to identify different types of sensitization. This facility is currently available only in select centers and is being conducted under research protocols.

In this study, we propose to: 1. evaluate the patterns of pain in CP and the triggers; 2. identify clinical surrogates of sensitization, i.e. neuropathic pain.

The ultimate goal is to apply the best possible pain management strategy based on our research findings for patients with CP in a personalised manner.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 years of disease (chronic pancreatitis)
* Both genders
* Able to provide informed consent

Exclusion Criteria:

* Acute exacerbation of chronic pancreatitis
* Moderate to severe abdominal pain at the time of screening
* Pancreatic cancer or other malignancies
* Use of antidepressants, narcotics, and neuromodulators

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with documented CP will be screened for enrolment criteria. Those fulfilling criteria will be enrolled after written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Type of pain | 18 months
  The type of pancreatic pain, i.e nociceptive or neuropathic will be determined
Quality of life | 18 months
  EORTC QLQ c30 score
Mental status | 18 months
  Depression and anxiety will be determined
Neural sensitization | 18 months
  Presence of localised and widespread sensitisation will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Drewes AM, Bouwense SAW, Campbell CM, Ceyhan GO, Delhaye M, Demir IE, Garg PK, van Goor H, Halloran C, Isaji S, Neoptolemos JP, Olesen SS, Palermo T, Pasricha PJ, Sheel A, Shimosegawa T, Szigethy E, Whitcomb DC, Yadav D; Working group for the International (IAP - APA - JPS - EPC) Consensus Guidelines for Chronic Pancreatitis. Guidelines for the understanding and management of pain in chronic pancreatitis. Pancreatology. 2017 Sep-Oct;17(5):720-731. doi: 10.1016/j.pan.2017.07.006. Epub 2017 Jul 13. PMID 28734722
- [Background] Faghih M, Phillips AE, Kuhlmann L, Afghani E, Drewes AM, Yadav D, Singh VK, Olesen SS; Pancreatic Quantitative Sensory Testing (P-QST) Consortium. Pancreatic QST Differentiates Chronic Pancreatitis Patients into Distinct Pain Phenotypes Independent of Psychiatric Comorbidities. Clin Gastroenterol Hepatol. 2022 Jan;20(1):153-161.e2. doi: 10.1016/j.cgh.2020.10.036. Epub 2020 Oct 22. PMID 34108130
- [Background] Talukdar R, Reddy DN. Pain in chronic pancreatitis: managing beyond the pancreatic duct. World J Gastroenterol. 2013 Oct 14;19(38):6319-28. doi: 10.3748/wjg.v19.i38.6319. PMID 24151350
- [Background] Sarkar S, Sarkar P, M R, Hazarika D, Prasanna A, Pandol SJ, Unnisa M, Jakkampudi A, Bedarkar AP, Dhagudu N, Reddy DN, Talukdar R. Pain, depression, and poor quality of life in chronic pancreatitis: Relationship with altered brain metabolites. Pancreatology. 2022 Sep;22(6):688-697. doi: 10.1016/j.pan.2022.06.007. Epub 2022 Jun 8. PMID 35710761